CLINICAL TRIAL: NCT02143310
Title: A Multi-Centre Study to Evaluate the Safety of Use of Electronic Vapour Products for Two Years
Brief Title: A Study to Evaluate the Safety of Electronic Vapor Products for 2 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fontem Ventures BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EVP G1 S3
Record Dates: First submitted 2014-05-09; First posted 2014-05-21 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EVP (Experimental): Subject who use the EVP for up to 2 years
  Interventions: Device: EVP

INTERVENTIONS:
Device: EVP

SUMMARY:
Electronic Vapour Products (EVPs) is a relatively new class of consumer products that are otherwise known as electronic cigarettes devices/systems. These may look like conventional cigarettes but do not contain tobacco.

The 'vapour' produced by such devices typically consists of humectants (propylene glycol or glycerol), nicotine, water, and flavours.

This trial is to evaluate the safety and tolerability of an EVP over two years.

ELIGIBILITY:
Inclusion Criteria:

* Subject who participated in the EVP G1 S2 study (S2)
* Willingness to use the EVP provided by the sponsor for two years as the only nicotine containing product
* No clinically significant abnormalities during the S2 study

Exclusion Criteria:

* Subjects who have used nicotine replacement therapy during the S2 study
* Subjects with relevant illness history
* Subjects with history of drug or alcohol abuse
* Subjects with lung function test or vital signs considered unsuitable Subjects who are trying to stop smoking
* Female subjects who are pregnant, or unwilling to use acceptable contraceptive method for the duration of the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12-29 (Actual); Study Completion 2016-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MD, Principal Investigator — Covance Clinical Research Unit
Locations (2):
- United Kingdom (2):
  - Covance Clinical Research Unit, Leeds, England
  - Simbec Research, Merthyr Tydfil, Wales

RESULTS

PARTICIPANT FLOW:
Groups:
- EVP Users: Subject who switch to use the electronic vapour product (EVP) for up to 2 years
  EVP
Period: Overall Study
Arm/Group | EVP Users
Started | 209
Completed | 102
Not Completed | 107

BASELINE CHARACTERISTICS:
Groups:
- EVP Users: Subjects who switch to use the EVP for up to 2 years
  EVP
Arm/Group | EVP Users
Number analyzed (Participants) | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 115
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Exhaled carbon monoxide (CO) [Mean (Standard Deviation); unit: ppm] | 13.6 (11.1)
Carboxyhemoglobin [Mean (Standard Deviation); unit: Percent of total hemoglobin] | 5.09 (2.04)
HDL cholesterol [Mean (Inter-Quartile Range); unit: mmol/L] — High density lipoprotein (HDL) cholesterol, in mmol/L
  mmol/L | 1.41 [1.35 to 1.46]
Biomarkers of exposure to nicotine [Mean (Standard Deviation); unit: mg] — The baseline amount of nicotine equivalents excreted in urine in 24-hours (AE24h).
  mg | 8.39 (7.19)
Level of white blood cells [Mean (Inter-Quartile Range); unit: G/L] | 7.3 [7.05 to 7.55]

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure
Description: Sitting systolic blood pressure (mmHg)
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- EVP Users: Subjects who use the EVP
  EVP
Arm/Group | EVP Users
Number analyzed (Participants) | 102
mmHg | 122.4 (11.1)

2. Primary Outcome: Electrocardiogram (ECG): PR Interval
Description: In electrocardiography, the PR interval is the period that extends from the beginning of the P wave (the onset of atrial depolarization) until the beginning of the QRS complex. Variations in the PR interval can be associated with certain medical conditions.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | EVP Users
Number analyzed (Participants) | 102
ms | 152.3 (18.7)

3. Primary Outcome: Lung Function Tests
Description: Forced Vital Capacity (FVC)
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | EVP Users
Number analyzed (Participants) | 102
Liters | 4.369 (1.007)

4. Primary Outcome: Clinical Laboratory Parameters
Description: High density lipoprotein (HDL) cholesterol, change from baseline (BL)
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | EVP Users
Number analyzed (Participants) | 102
mmol/L | -0.03 [-0.08 to 0.02]

5. Secondary Outcome: Nicotine Withdrawal Symptoms
Description: Nicotine withdrawal symptoms were measured using the revised Minnesota Nicotine Withdrawal Scale (MWS-R) questionnaire. Extended total scores were used, i.e. the sum of the scores of all 15 questions of the questionnaire. Symptoms (e.g. angry, irritable, frustrated, depressed, restless, insomnia) were rated from 0 (none) to 4 (severe). Extended total scores may range from 0 to a maximum of 60.
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EVP Users
Number analyzed (Participants) | 102
score on a scale | 3.3 (4.2)

6. Secondary Outcome: Biomarkers of Exposure to Nicotine
Description: The exposure to nicotine was measured by quantifying the change from BL in the amount of nicotine equivalents excreted in urine in 24-hours (AE24h).
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | EVP Users
Number analyzed (Participants) | 102
mg | 0.85 [-0.17 to 1.88]

7. Secondary Outcome: Biomarkers of Effect
Description: Change from BL in the level of white blood cells.
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: G/L
Arm/Group | EVP Users
Number analyzed (Participants) | 102
G/L | -0.31 [-0.62 to 0.00]

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | EVP Users
All-Cause Mortality (participants affected / at risk) | 0/209
Serious Adverse Events (participants affected / at risk) | 7/209
Other Adverse Events (participants affected / at risk) | 60/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EVP Users (N=209)
Acute pancreatitis (Gastrointestinal disorders) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Right occipital stroke (Nervous system disorders) | 1
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 2
Pneumonia (Infections and infestations) | 1
Joint injury (Injury, poisoning and procedural complications) | 1 — Right knee injury
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EVP Users (N=209)
Headache (Nervous system disorders) | 60
Nasopharyngitis (Infections and infestations) | 60
Influenza (Infections and infestations) | 18
Urinary tract infection (Infections and infestations) | 12
Sore throat (Respiratory, thoracic and mediastinal disorders) | 41
Cough (Respiratory, thoracic and mediastinal disorders) | 35
Nicotine dependence (Psychiatric disorders) | 25
Toothache (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 15
Seasonal allergy (Immune system disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No